CLINICAL TRIAL: NCT02634580
Title: A Double-blind, Randomized, Multicenter Study to Evaluate the Safety and Efficacy of Evolocumab, Compared With Ezetimibe, in Hypercholesterolemic Japanese Subjects Unable to Tolerate an Effective Dose of a HMG-CoA Reductase Inhibitor Due to Muscle Related Side Effects
Brief Title: Goal Achievement After Utilizing an Anti-PCSK9 Antibody in Statin Intolerant Subjects-4
Acronym: GAUSS-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20140234
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Hypercholesterolemia
Keywords: Japanese; High cholesterol; Treatment of high cholesterol; Lowering cholesterol; Lowering high cholesterol; Hypercholesterolemia; Statin intolerant
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ezetimibe (Q2W) (Active Comparator): Participants received placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe orally once a day for 12 weeks. From week 12 participants received open-label evolocumab 140 mg subcutaneously once every 2 weeks until week 48.
  Interventions: Biological: Evolocumab; Drug: Ezetimibe; Drug: Placebo to Evolocumab
- Ezetimibe (QM) (Active Comparator): Participants received placebo subcutaneous injection once a month and 10 mg ezetimibe orally once a day for 12 weeks. From week 12 participants received open-label evolocumab 420 mg subcutaneously once a month until week 48.
  Interventions: Biological: Evolocumab; Drug: Ezetimibe; Drug: Placebo to Evolocumab
- Evolocumab Q2W (Experimental): Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks and placebo tablets once a day for 12 weeks. From week 12 participants received open-label evolocumab 140 mg subcutaneously once every 2 weeks until week 48.
  Interventions: Biological: Evolocumab; Drug: Placebo Ezetimibe
- Evolocumab QM (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once a day for 12 weeks. From week 12 participants received open-label evolocumab 420 mg subcutaneously once a month until week 48.
  Interventions: Biological: Evolocumab; Drug: Placebo Ezetimibe

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
Drug: Ezetimibe — Tablet for oral administration
  Other Names: Zetia
  Arms: Ezetimibe (Q2W); Ezetimibe (QM)
Drug: Placebo to Evolocumab — Administered by subcutaneous injection
  Arms: Ezetimibe (Q2W); Ezetimibe (QM)
Drug: Placebo Ezetimibe — Tablet for oral administration
  Arms: Evolocumab Q2W; Evolocumab QM

SUMMARY:
The primary objective of the study was to evaluate the effect of 12 weeks of subcutaneous (SC) evolocumab compared with ezetimibe, on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) in hypercholesterolemic adults unable to tolerate an effective dose of a statin.

DETAILED DESCRIPTION:
After screening participants who met all inclusion/exclusion criteria were randomized with an allocation ratio of 2:2:1:1 into 4 groups: evolocumab (AMG 145) 420 mg administered by subcutaneous injection monthly and placebo pill daily; evolocumab 140 mg administered by subcutaneous injection every two weeks and placebo pill by mouth daily; placebo 420 mg administered by subcutaneous injection monthly and ezetimibe 10 mg pill daily; placebo 140 mg administered subcutaneous injection every two weeks and ezetimibe 10 mg pill daily. Randomization was stratified by screening LDL-C level and baseline statin use. Participants on low or atypical statin dose therapy must have been on a stable dose for at least 4 weeks prior to screening and throughout the blinded portion of the study; the dose could not be adjusted during screening and for the duration of the study. After Week 12, ezetimibe was discontinued and participants moved to an open-label dose of evolocumab administered by subcutaneous injection either every two weeks or monthly and their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 20 to ≤ 80 years of age
* Japanese by self-identification
* Not on a statin or on a low dose statin with stable dose for at least 4 weeks.
* Subject not at LDL-C goal
* History of statin intolerance to at least 2 statins
* Lipid lowering therapy has been stable prior to screening for at least 4 weeks
* Fasting triglycerides ≤ 400 mg/dL

Exclusion Criteria:

* New York Heart Association (NYHA) III or IV heart failure
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Type 1 diabetes
* Poorly controlled type 2 diabetes
* Uncontrolled hypothyroidism or hyperthyroidism

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-02-27 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2018-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- Japan (30):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Chiba, Chiba
  - Research Site, Kisarazu-shi, Chiba
  - Research Site, Matsudo-shi, Chiba
  - Research Site, Chikushino-shi, Fukuoka
  - Research Site, Koga-shi, Fukuoka
  - Research Site, Sukagawa-shi, Fukushima
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Kobe, Hyōgo
  - Research Site, Koga-shi, Ibaraki
  - Research Site, Kahoku-gun, Ishikawa-ken
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Komatsu-shi, Ishikawa-ken
  - Research Site, Morioka, Iwate
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Ohsaki-shi, Miyagi
  - Research Site, Nakagami-gun, Okinawa
  - Research Site, Osaka, Osaka
  - Research Site, Fujimi-shi, Saitama
  - Research Site, Iruma-gun, Saitama
  - Research Site, Kawaguchi-shi, Saitama
  - Research Site, Hamamatsu, Shizuoka
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Higashiyamato-shi, Tokyo
  - Research Site, Musashino-shi, Tokyo
  - Research Site, Shinagawa-ku, Tokyo

REFERENCES:
- [Derived] Koba S, Inoue I, Cyrille M, Lu C, Inomata H, Shimauchi J, Kajinami K. Evolocumab vs. Ezetimibe in Statin-Intolerant Hyperlipidemic Japanese Patients: Phase 3 GAUSS-4 Trial. J Atheroscler Thromb. 2020 May 1;27(5):471-484. doi: 10.5551/jat.50963. Epub 2019 Nov 21. PMID 31748467
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 30 centers in Japan. Participants were enrolled from 27 February 2016 to 18 May 2017.
  The study consisted of a 12-week double-blind (DB) treatment period and a 9-month open-label extension (OLE) period.
Pre-assignment Details: Participants were randomized 1:1:2:2 into 1 of 4 treatment groups for the 12-week, double-blind treatment period. Randomization was stratified by screening low-density lipoprotein cholesterol (LDL-C) level (< 180 mg/dL vs. ≥ 180 mg/dL) and baseline statin use (yes vs. no).
Groups:
- Ezetimibe (Q2W): Participants received placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe orally once a day for 12 weeks in the double-blind treatment period.
  From week 12 to week 48 participants self-administered 140 mg evolocumab subcutaneously every 2 weeks in the open-label extension period.
- Ezetimibe (QM): Participants received placebo subcutaneous injection once a month and 10 mg ezetimibe orally once a day for 12 weeks in the double-blind treatment period.
  From week 12 to week 48 participants self-administered 420 mg evolocumab subcutaneously once a month in the open-label extension period.
- Evolocumab Q2W: Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks and placebo tablets once a day for 12 weeks in the double-blind treatment period.
  From week 12 to week 48 participants self-administered 140 mg evolocumab subcutaneously every 2 weeks in the open-label extension period.
- Evolocumab QM: Participants received 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once a day for 12 weeks in the double-blind treatment period.
  From week 12 to week 48 participants self-administered 420 mg evolocumab subcutaneously once a month in the open-label extension period.
Period: Double-blind Treatment Period
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Started | 10 | 11 | 19 | 21
Completed (Completed double-blind treatment period) | 9 | 11 | 18 | 20
Not Completed | 1 | 0 | 1 | 1
Not completed — Subject Request | 1 | 0 | 1 | 1
Period: Open-label Extension Period
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM
Started | 9 | 11 | 18 | 21 (Includes 1 participant who did not complete the double-blind period but had study visits during OLE)
Received Open-label Treatment | 9 | 11 | 18 | 20
Completed (Completed study) | 9 | 10 | 18 | 20
Not Completed | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ezetimibe (Q2W): Participants received placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe orally once a day for 12 weeks.
- Ezetimibe (QM): Participants received placebo subcutaneous injection once a month and 10 mg ezetimibe orally once a day for 12 weeks.
- Evolocumab Q2W: Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks and placebo tablets once a day for 12 weeks.
- Evolocumab QM: Participants received 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once a day for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Ezetimibe (Q2W) | Ezetimibe (QM) | Evolocumab Q2W | Evolocumab QM | Total
Number analyzed (Participants) | 10 | 11 | 19 | 21 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.8) | 58.7 (12.5) | 65.1 (10.5) | 66.4 (9.3) | 64.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 9 | 12 | 31
  Male | 5 | 6 | 10 | 9 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 10 | 11 | 19 | 21 | 61
Intolerance to Statins [Count of Participants; unit: Participants]
  One statin | 1 | 0 | 1 | 0 | 2
  Two statins | 7 | 10 | 14 | 14 | 45
  Three statins | 2 | 1 | 3 | 4 | 10
  Four or more statins | 0 | 0 | 1 | 3 | 4
Stratification Factor: Screening LDL-C Level [Count of Participants; unit: Participants]
  < 180 mg/dL [4.66 mmol/L] | 5 | 6 | 9 | 10 | 30
  ≥ 180 mg/dL [4.66 mmol/L] | 5 | 5 | 10 | 11 | 31
Stratification Factor: Baseline Statin Use [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 3 | 5 | 14
  No | 7 | 8 | 16 | 16 | 47
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] | 181.0 (34.7) | 182.7 (72.2) | 198.1 (64.1) | 188.0 (41.6) | 189.0 (53.9)
Total Cholesterol Concentration [Mean (Standard Deviation); unit: mg/dL] | 280.0 (34.4) | 275.2 (79.7) | 282.0 (63.9) | 282.3 (49.6) | 280.5 (57.3)
High-density Lipoprotein Cholesterol (HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 62.5 (15.6) | 64.1 (16.1) | 54.3 (18.2) | 64.1 (20.9) | 60.8 (18.6)
Very Low-density Lipoprotein Cholesterol (VLDL) Concentration [Mean (Standard Deviation); unit: mg/dL] | 36.5 (21.9) | 28.4 (16.1) | 29.6 (12.0) | 30.2 (12.3) | 30.7 (14.7)
Triglycerides Concentration [Mean (Standard Deviation); unit: mg/dL] | 183.1 (111.1) | 142.3 (80.1) | 148.0 (59.8) | 151.0 (61.3) | 153.8 (73.7)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 132.1 (19.4) | 121.9 (29.3) | 140.4 (31.7) | 138.7 (26.2) | 135.1 (27.9)
Non-HDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] | 217.5 (37.3) | 211.1 (71.2) | 227.7 (63.3) | 218.2 (42.2) | 219.8 (53.7)
Total cholesterol/HDL-C ratio [Mean (Standard Deviation); unit: ratio] | 4.8 (1.4) | 4.4 (1.1) | 5.7 (2.0) | 4.8 (1.4) | 5.0 (1.6)
ApolipoproteinB/Apolipoprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] | 0.8 (0.2) | 0.8 (0.2) | 1.0 (0.4) | 0.9 (0.2) | 0.9 (0.3)
Lipoprotein(a) Concentration [Mean (Standard Deviation); unit: nmol/L] | 48.0 (72.3) | 66.0 (83.2) | 61.3 (72.6) | 66.2 (91.0) | 61.7 (79.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at the Mean of Weeks 10 and 12
Description: For all efficacy endpoints the two dosing regimens (every 2 weeks and every month) for each treatment were pooled for analysis.
Time Frame: Baseline and Weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Ezetimibe: Participants received placebo subcutaneous injection once every 2 weeks or once a month and 10 mg ezetimibe orally once a day for 12 weeks.
- Evolocumab: Participants received SC evolocumab 140 mg once every 2 weeks or 420 mg once a month and placebo tablets once a day for 12 weeks.
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -20.39 (3.19) | -59.75 (2.30)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Model includes treatment group, stratification factor (screening LDL-C level), scheduled visit and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -39.35, 95% CI 2-sided [-47.23 to -31.48], Standard Error of Mean 3.93 — Evolocumab - Ezetimibe

2. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -19.13 (3.45) | -59.27 (2.50)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -40.14, 95% CI 2-sided [-48.68 to -31.60], Standard Error of Mean 4.26 — Evolocumab - Ezetimibe

3. Secondary Outcome: Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
mg/dL | -35.6 (6.6) | -113.2 (4.8)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -77.6, 95% CI 2-sided [-93.9 to -61.3], Standard Error of Mean 8.1 — Evolocumab - Ezetimibe

4. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
mg/dL | -33.4 (7.0) | -112.7 (5.1)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -79.4, 95% CI 2-sided [-96.7 to -62.0], Standard Error of Mean 8.7 — Evolocumab - Ezetimibe

5. Secondary Outcome: Percentage of Participants Who Achieved a Mean LDL-C at Weeks 10 and 12 of Less Than 70 mg/dL
Description: Mean low density lipoprotein-cholesterol response was defined as LDL-C < 70 mg/dL [1.8 mol/L].
Time Frame: Weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percentage of participants | 0.00 [0.00 to 16.11] | 56.41 [40.98 to 70.70]
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran Mantel Haenszel (CMH) test adjusted by the stratification factor (screening LDL-C level); Treatment Difference = 56.41, 95% CI 2-sided [34.10 to 70.70] — Evolocumab - Ezetimibe

6. Secondary Outcome: Percentage of Participants Who Achieved a LDL-C of Less Than 70 mg/dL at Week 12
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percentage of participants | 0.00 [0.00 to 16.11] | 52.63 [37.26 to 67.52]
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran Mantel Haenszel (CMH) test adjusted by the stratification factor (screening LDL-C level); Treatment Difference = 52.63, 95% CI 2-sided [30.36 to 67.52] — Evolocumab - Ezetimibe

7. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -13.80 (2.17) | -39.24 (1.57)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -25.44, 95% CI 2-sided [-30.80 to -20.08], Standard Error of Mean 2.68 — Evolocumab - Ezetimibe

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -12.69 (2.34) | -38.52 (1.70)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -25.83, 95% CI 2-sided [-31.63 to -20.04], Standard Error of Mean 2.89 — Evolocumab - Ezetimibe

9. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -18.82 (2.77) | -52.35 (2.01)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.53, 95% CI 2-sided [-40.38 to -26.68], Standard Error of Mean 3.42 — Evolocumab - Ezetimibe

10. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -18.28 (3.03) | -51.71 (2.20)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.44, 95% CI 2-sided [-40.94 to -25.94], Standard Error of Mean 3.75 — Evolocumab - Ezetimibe

11. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -13.23 (2.69) | -48.90 (1.93)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -35.67, 95% CI 2-sided [-42.30 to -29.04], Standard Error of Mean 3.31 — Evolocumab - Ezetimibe

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -11.32 (2.99) | -47.91 (2.14)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -36.60, 95% CI 2-sided [-43.98 to -29.22], Standard Error of Mean 3.68 — Evolocumab - Ezetimibe

13. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -15.73 (2.69) | -44.34 (1.94)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.61, 95% CI 2-sided [-35.26 to -21.97], Standard Error of Mean 3.32 — Evolocumab - Ezetimibe

14. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -17.34 (2.81) | -44.39 (2.04)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.05, 95% CI 2-sided [-34.00 to -20.09], Standard Error of Mean 3.47 — Evolocumab - Ezetimibe

15. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A-1 Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -15.39 (2.67) | -52.46 (1.91)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -37.07, 95% CI 2-sided [-43.65 to -30.50], Standard Error of Mean 3.28 — Evolocumab - Ezetimibe

16. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A-1 Ratio at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -15.62 (2.88) | -51.91 (2.06)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -36.29, 95% CI 2-sided [-43.39 to -29.20], Standard Error of Mean 3.54 — Evolocumab - Ezetimibe

17. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -5.89 (4.34) | -37.02 (3.11)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.13, 95% CI 2-sided [-41.83 to -20.43], Standard Error of Mean 5.34 — Evolocumab - Ezetimibe

18. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -5.21 (5.02) | -36.41 (3.59)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.21, 95% CI 2-sided [-43.57 to -18.84], Standard Error of Mean 6.17 — Evolocumab - Ezetimibe

19. Secondary Outcome: Percent Change From Baseline in Triglycerides at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -5.21 (5.92) | -1.73 (4.28)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.63, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 3.49, 95% CI 2-sided [-11.15 to 18.13], Standard Error of Mean 7.31 — Evolocumab - Ezetimibe

20. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -9.87 (7.71) | 1.92 (5.60)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.22, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 11.79, 95% CI 2-sided [-7.29 to 30.87], Standard Error of Mean 9.52 — Evolocumab - Ezetimibe

21. Secondary Outcome: Percent Change From Baseline in HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | 3.10 (2.50) | 11.06 (1.80)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.012, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 7.96, 95% CI 2-sided [1.78 to 14.14], Standard Error of Mean 3.08 — Evolocumab - Ezetimibe

22. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | 6.45 (2.59) | 12.04 (1.88)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.086, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 5.59, 95% CI 2-sided [-0.82 to 12.00], Standard Error of Mean 3.20 — Evolocumab - Ezetimibe

23. Secondary Outcome: Percent Change From Baseline in VLDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -4.67 (5.89) | -5.34 (4.25)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.93, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -0.67, 95% CI 2-sided [-15.22 to 13.87], Standard Error of Mean 7.26 — Evolocumab - Ezetimibe

24. Secondary Outcome: Percent Change From Baseline in VLDL-C at Week 12
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 21 | 40
percent change | -9.06 (8.00) | -1.42 (5.80)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.44, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 7.64, 95% CI 2-sided [-12.15 to 27.43], Standard Error of Mean 9.88 — Evolocumab - Ezetimibe

ADVERSE EVENTS:
Time Frame: Double-blind Treatment Period: From randomization (for all-cause mortality) or first dose of study drug (for adverse events) up to week 12 or the day before OLE day 1. Open-label Extension Period: From the start of the OLE (week 12) to end of study (week 54) for all-cause mortality (up to 42 weeks); and from first dose of study drug in the OLE up to 30 days after last dose, or end of study, whichever was earlier, for adverse events (a maximum of 40 weeks).
Description: Adverse events are reported for all participants who received at least one dose of study drug in each period. All-cause mortality is reported for all participants randomized in the double-blind treatment period and for all participants who entered the OLE period.
Groups:
- DB Period: Ezetimibe (Q2W): Participants received placebo subcutaneous injection once every 2 weeks and 10 mg ezetimibe orally once a day for 12 weeks.
- DB Period: Ezetimibe (QM): Participants received placebo subcutaneous injection once a month and 10 mg ezetimibe orally once a day for 12 weeks.
- DB Period: Evolocumab Q2W: Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks and placebo tablets once a day for 12 weeks.
- DB Period: Evolocumab QM: Participants received 420 mg evolocumab by subcutaneous injection once a month and placebo tablets once a day for 12 weeks.
- OLE Period: Evolocumab: Participants received evolocumab by subcutaneous injection from week 12 to week 48 at the same dosing interval as the investigational product regimen that they were randomized to during the double-blind period (ie, every 2 weeks or once monthly) during the open-label extension (OLE) period.
Arm/Group | DB Period: Ezetimibe (Q2W) | DB Period: Ezetimibe (QM) | DB Period: Evolocumab Q2W | DB Period: Evolocumab QM | OLE Period: Evolocumab
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/19 | 0/21 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/11 | 0/19 | 0/21 | 4/58
Other Adverse Events (participants affected / at risk) | 4/10 | 8/11 | 11/19 | 12/21 | 44/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Ezetimibe (Q2W) (N=10) | DB Period: Ezetimibe (QM) (N=11) | DB Period: Evolocumab Q2W (N=19) | DB Period: Evolocumab QM (N=21) | OLE Period: Evolocumab (N=58)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Ezetimibe (Q2W) (N=10) | DB Period: Ezetimibe (QM) (N=11) | DB Period: Evolocumab Q2W (N=19) | DB Period: Evolocumab QM (N=21) | OLE Period: Evolocumab (N=58)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral mucosa haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 2 | 1
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 5 | 17
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 1 | 2
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Onychomalacia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 3
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT02634580/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT02634580/SAP_001.pdf